CLINICAL TRIAL: NCT03450668
Title: Comparison of the mOm Incubator With a Standard Incubator for the Maintenance of Thermal Stability in Preterm Infants With User Feedback
Brief Title: mOm Incubator Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: mOm incubators (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Supportive Care
Other Study IDs: mOm/2018/01
Record Dates: First submitted 2018-02-23; First posted 2018-03-01 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Hypothermia
Keywords: neonatal, incubator, thermal-regulation
MeSH Terms: conditions — Hypothermia

STUDY DESIGN:
Intervention Model Description: a randomized two-arm crossover study
Who Masked: Participant, Care Provider, Investigator
Masking Description: Choice of incubator used is randomized and blinded until the subject has been recruited and incubator arm assigned. After which it will be known to all concerned.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- standard incubator (Active Comparator): routinely used standard incubator already used in the neonatal unit
  Interventions: Device: mOm incubator; Device: standard incubator
- mOm incubator (Experimental): new test incubator
  Interventions: Device: mOm incubator; Device: standard incubator

INTERVENTIONS:
Device: mOm incubator — 24 hour usage of test incubator
Device: standard incubator — standard incubator

SUMMARY:
The mOm Incubator is a collapsible infant incubator designed to provide a level of thermoregulation that meets the standards set for conventional incubators whilst being low cost and space-saving. Babies recruited will be clinically stable, at least 30 weeks gestational age and require at least 48 hours incubator care. A standard or test incubator will be used for the first 24 hours chosen randomly, then the baby will be moved to the over arm for a further 24 hours.

DETAILED DESCRIPTION:
Investigators will recruit babies who are in the Neonatal Unit at St. Peter's Hospital. Babies will be clinically stable from a cardio-respiratory point of view. They will also be requiring incubator care (so they will weigh less than approximately 1400g) but not requiring additional humidification. This effectively excludes babies born less than 30 weeks gestation who are routinely humidified for the first week (if 28-30 weeks gestation) or two weeks (if less than 28 weeks gestation). Some term babies may also be eligible for the study if they are being nursed in an incubator for clinical reasons.

Identification and recruitment of babies will be carried out by the attending Consultant Neonatologist and the research team.

For twins, consecutive enrolment will be possible if only one mOm incubator is available.

There will be two arms to the protocol. The first arm will consist of standard incubator care, where the care of the baby is unchanged, but non-invasive, more frequent (hourly) temperature and other physiological measures of stability than would normally be collected in routine care (nominally every three hours) will be collected. The second arm will be the baby receiving normal care in the mOm incubator, with another set of hourly detailed, non-invasive, observations. The planned care and monitoring of the baby will be otherwise unchanged. No additional blood tests or any other invasive testing or monitoring are required. The clinical team will have full control and responsibility for the baby's care and can terminate the study for the baby at any time for any reason.

In addition, investigators will collect the views of staff on the baby's comfort, visibility, care, usability and acceptability during each arm of the study.

For each arm of the study, the secondary outcome measures are:

(1) pulse rate (as a measure of clinical stability) (2) respiratory rate (as a measure of clinical stability) (3) apnea and bradycardia episodes recorded by nursing staff (clinical stability) (4) temperature (as a measure of clinical stability) (4) adverse events related to incubator performance (5) cleaning ease and time took (6) set up time (7) staff structured feedback

36 eligible babies will be recruited into the study at a single site, being identified by the clinical team. All 36 will experience a 24 hour period in each of the two incubators (mOm and standard) (48 hours in total), in a randomly allocated order. Babies will act as their own controls in this cross-over study design. If any babies fail to complete the 48-hour study procedures (e.g. due to data incomplete or baby withdrawn) further babies will be recruited to achieve 36 complete datasets.

ELIGIBILITY:
Inclusion Criteria:

* At least 30 weeks gestational age and less than or equal to 6kg
* In need of at least 48 hours incubation in a stable temperature environment
* Must be clinically stable
* Parental/legal guardian written informed consent has been given

Exclusion Criteria:

* Does not require humidity regulation
* Parent/legal guardian must not be from a vulnerable group

Ages: 1 Minute to 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 74 (Actual)
Dates: Start 2021-10-27 (Actual); Primary Completion 2022-08-04 (Actual); Study Completion 2022-08-04 (Actual)

PRIMARY OUTCOMES:
thermo-regulation | 24 hours
  ability of incubator to maintain stable temperature of baby

SECONDARY OUTCOMES:
Usability | 24 hours
  Time to prepare for use and clean incubator (in-use cleaning and deep clean between use)

CONTACTS AND LOCATIONS:
Locations (1):
- Ashford and St. Peter's Hospital, Chertsey, Surrey, United Kingdom

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2022-03-09): https://cdn.clinicaltrials.gov/large-docs/68/NCT03450668/Prot_SAP_ICF_000.pdf